CLINICAL TRIAL: NCT03129607
Title: An Observational Retrospective Study in Postoperative Pancreatic Fistula
Brief Title: A Study in Postoperative Pancreatic Fistula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZhejiangU06
Record Dates: First submitted 2017-04-04; First posted 2017-04-26 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
Keywords: POPF; Classification system
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POPF group: Patients who had POPF will be included into POPF group.
- Observation group: Patients without POPF will be included into observation group.

SUMMARY:
The International Study Group of Pancreatic Surgery (ISGPS) issued the definition and classification system of postoperative pancreatic fistula (POPF), and received widespread recognition. Currently, it has become an important reference for clinical treatment of POPF.

DETAILED DESCRIPTION:
The definition of POPF released by ISGPS in 2016 still seems to have certain deficiency. For example, in both definitions in 2005 and 2016, the re-operation is used as an important judgment index of "Grade C POPF". But a unified standard or consensus is still lacked for the indication of POPF re-operation, which may finally impact the diagnosis of "Grade C POPF". Therefore, we performed this study, so as to better improve the relevant definition and provide guidance for the diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of POPF;
* Aged 18 or older;
* Of either sex.

Exclusion Criteria:

* No specific exclusion criteria will be applied to a participant as long as the participant is eligible for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosed POPF
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic fistula | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 200 days
  The determine of pancreatic fistula follows the International Study Group on Pancreatic Fistulas (ISGPF) criteria

SECONDARY OUTCOMES:
Hospital stays | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 200 days
  Post-operation hospital stay is assessed
Number of hospitalizations | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 200 days
  Number of hospitalizations during the observational period
Mortality | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 200 days
  Postoperative death in 30 days are considered concerned with pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Bo Liang, phD, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No